CLINICAL TRIAL: NCT01131988
Title: An Open Label, Two Way Crossover, Balanced, Single Dose, Comparative Evaluation of Relative Bioavailability of Tacrolimus Capsules 5 mg With That of 'Prograf' Capsules 5 mg in Healthy Subjects Under Fasting Conditions.
Brief Title: Bioavailability Study of Tacrolimus Capsules, 5 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. Ramesh Mullangi/Director - R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA0859002
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioavailability, crossover, tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Experimental): Tacrolimus Capsules, 5 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Tacrolimus Capsules
- Prograf Capsules (Active Comparator): Prograf Capsules of Astellas Pharma US, Inc.,
  Interventions: Drug: Tacrolimus Capsules

INTERVENTIONS:
Drug: Tacrolimus Capsules — Tacrolimus Capsules, 5 mg of Dr. Reddy's Laboratories Limited
  Other Names: Prograf capsules of Astellas Pharma US, Inc.,

SUMMARY:
The purpose of this study is to compare the relative bioavailability study of tacrolimus capsules 5 mg with prograf capsules 5 mg in healthy, adult, human subjects under fasting conditions and to monitor safety of subjects

DETAILED DESCRIPTION:
An open label, randomized, two period, two treatment, two sequence, crossover, balanced, single dose, comparative evaluation of relative bioavailability of tacrolimus capsules 5 mg with that of 'prograf' capsules 5 mg in healthy adult human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be healthy human between 18 and 45 years.
2. The subjects should be screened within 21 days prior to the administration of first dose of the study drug.
3. The subjects should have a BMI between 18.5 and 24.9 weight in kg/ height2 in meter.
4. The subjects should be able to communicate effectively with study personnel.
5. The subjects should be able to give written informed consent to participate in the study.

   If subject is a female volunteer and
6. Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms,foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
7. Is postmenopausal for at least 1 year.
8. Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. The subjects who have a history of allergic responses to tacrolimus or other related drugs.
2. The subjects who have significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG, and X-ray recordings.
3. The subjects who have any disease or condition which might compromise the haemopoeitic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
4. The subjects who have a history or presence of bronchial asthma.
5. The subjects who have used enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
6. The subjects who have history of drug dependence, recent history of alcoholism or of moderate alcohol uses.
7. The subjects who are smokers who smoke more than or equal to 10 cigarettes per day or more than or equal to 20 biddies per day or those who cannot refrain from smoking during study period.
8. The subjects with a history of difficulty with donating blood or difficulty in accessibility of veins.
9. The subjects who have donated 1 unit (350 ml / 450 ml) blood within 90 days prior to receiving the first dose of study medication.
10. The subjects who have a positive hepatitis screen (include subtypes A, B, C and E).
11. The subjects who have a positive test result for HIV antibody and / or syphilis (RPR/VDRL).
12. The subject who receives an investigational product, or has participated in a drug research study within a period of 90 days prior to the first dose of the study medication application.
13. Female volunteers demonstrating a positive pregnancy screen.
14. Female volunteers who are currently breast-feeding.
15. Female volunteers not willing to use contraception during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability study based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Simran Sethi, MBBS, Principal Investigator — BA Research India Limited
Locations (1):
- BA Research India Limited, Ahmedabad, Gujarat, India